CLINICAL TRIAL: NCT00572832
Title: Randomized Trial of Alternative Quadrivalent Human Papilloma Virus (HPV) Vaccination Schedules in a University Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Richard K. Zimmerman, MD/Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 32090
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Results first posted 2010-02-25 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Human Papillomavirus Infection
Keywords: Human Papillomavirus Vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 mon. 3rd dose of quadrivalent human papillomavirus vaccine (Active Comparator): Receipt of three doses of quadrivalent human papillomavirus vaccine according to the regular schedule of 0,2, and 6 months.
  Interventions: Biological: Quadrivalent human papillomavirus vaccine on-time administration
- 12 mon. 3rd dose of quadrivalent human papillomavirus vaccine (Active Comparator): Receipt of three doses of quadrivalent human papillomavirus vaccine on a delayed schedule of 0,2, and 12 months.
  Interventions: Biological: Quadrivalent human papillomavirus vaccine delayed administration

INTERVENTIONS:
Biological: Quadrivalent human papillomavirus vaccine on-time administration — The vaccine is given in three doses: Dose 1; dose 2 given 60 days later; dose 3 given six months after dose 1.
  Other Names: Gardasil
  Arms: 6 mon. 3rd dose of quadrivalent human papillomavirus vaccine
Biological: Quadrivalent human papillomavirus vaccine delayed administration — The vaccine is given in three doses: Dose 1; dose 2 given 60 days later; dose 3 given 12 months after dose 1.
  Other Names: Gardasil
  Arms: 12 mon. 3rd dose of quadrivalent human papillomavirus vaccine

SUMMARY:
This is a randomized, open label trial of HPV (human papilloma virus) vaccine, comparing an on-time administration of the third dose with delayed administration of the third dose. All participants would receive the first and second doses according to schedule. They would be randomized to either vaccine at 6 months or vaccine at 12 months.

Blood will be drawn for titers twice from all participants: pre-dose 1 and one month post third dose. We hypothesize that the GMTs in the test group (T) are non-inferior to the usual timing control group (C):

H0: δ ≤ -δ0 versus H1: δ > -δ0 where δ = log (GMTT )- log (GMTC) and δ0 is the pre-specified non-inferiority margin.

DETAILED DESCRIPTION:
The recommendations for HPV vaccine include catch-up of women 18 to 26 years old. Given that a large percentage of women in this age group are attending college, a good place to access them would be through the student health services on college campuses. However, the HPV vaccine schedule of 0, 2, and 6 months is likely to be difficult to implement in a college calendar year and the immunogenicity of alternative schedules is unknown. If the immunogenicity of an altered schedule is good, then higher vaccination rates may be achievable.

Aims:

1. Determine if delay in the third dose is immunologically non-inferior to the standard administration schedule (1 month post-dose 3).
2. Determine the side effect profile of a delayed third dose, in comparison to the standard schedule

ELIGIBILITY:
Inclusion Criteria:

* 18-23 year old college females who are planning to return to the university for the next fall semester.

Exclusion Criteria:

* Pregnancy or planned pregnancy.
* Prior receipt of HPV vaccine.
* Greater than four lifetime sexual partners.
* Immunosuppression.
* Anti-coagulant therapy.
* Breastfeeding.
* History of abnormal pap smear.
* Allergy to vaccine components.

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Zimmerman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Zimmerman RK, Nowalk MP, Lin CJ, Fox DE, Ko FS, Wettick E, Cost G, Hand L, Hayes J, Michaels M. Randomized trial of an alternate human papillomavirus vaccine administration schedule in college-aged women. J Womens Health (Larchmt). 2010 Aug;19(8):1441-7. doi: 10.1089/jwh.2009.1753. PMID 20629576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred young women from the university community who met the eligibility criteria were recruited at the Student Health Service.
Groups:
- 6 Month Standard Schedule: Receipt of three doses of quadrivalent human papillomavirus vaccine according to the regular schedule of 0,2, and 6 months.
- 12 Month Alternative Group: 12 month Alternative Schedule Group with 3 doses of quadrivalent vaccine at 0, 2, and 12 months
Period: Overall Study
Arm/Group | 6 Month Standard Schedule | 12 Month Alternative Group
Started | 100 | 100
Completed | 100 | 88
Not Completed | 0 | 12
Not completed — Lost to Follow-up | 0 | 11
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 Month Standard Schedule | 12 Month Alternative Group | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 200
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 20.3 (1.3) | 20.1 (1.4) | 20.2 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 83 | 89 | 172
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.2 (4.7) | 24.5 (5.1) | 24.3 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Antibody Titers Following the Third Dose of Human Papilloma Virus (HPV) Vaccine by Virus Type and by Administration Schedule
Description: Geomtric mean antibody titers were assessed 1 month following the third dose of human papilloma virus vaccine. Persons with baseline antibody titers that were positive to a particular type were deleted from the analysis for that particular type so that the outcome is excludes those with baseline positives (thus, sample size varies by type). Responses were compared between the two groups after dose 3 by type.
Time Frame: 1 month post-dose 3 (i.e., 7 months for standard schedule and 13 months for alternative schedule)
Population: The analysis was by intention to treat. Participants who had positive baseline antibody titers were excluded from further analyses only for the type(s) for which they were seropositive.
Measure: Geometric Mean (95% Confidence Interval); unit: milliMerck units per mL
Arm/Group | 6 Month Standard Schedule | 12 Month Alternative Group
Number analyzed (Participants) | 100 | 88
milliMerck units per mL
  Type 6 | 1894 [1564 to 2194] | 4221 [2930 to 5416]
  Type 11 | 1773 [1261 to 2252] | 5623 [3939 to 7208]
  Type 16 | 5534 [3875 to 7093] | 11832 [8165 to 15223]
  Type 18 | 1225 [1038 to 1396] | 2052 [1138 to 2959]
Statistical Analysis 1: Comparison: 6 Month Standard Schedule vs 12 Month Alternative Group; Non-inferiority tested against 1-sided null hypothesis (alpha=.025) that the post Dose 3 GMT ratio of the Alternate to Standard schedule was ≤ 0.5 for each HPV type; Test type: Non-Inferiority or Equivalence — The formula used for calculating sample size for the treatment arm (NT) is NT = (1 + 1/u) (Zα + Zβ)2 σ2 /[log (RGMC) -δ0] where u is the ratio of the size of the control and treatment arms, one sided alpha that is divided by 4, a non-inferiority margin (δ0 of natural log 0.5), the expected ratio of geometric mean concentrations RGMC set at 0.8, and a standard deviation of 1.26 (the largest for HPV-16). The calculated sample size for a power of 80% was 75 participants in each arm; p = .025, ANOVA — Non-inferiority was tested against a one-sided null hypothesis (alpha=.025) that the post Dose 3 GMT ratio of the Alternate to Standard schedule was ≤ 0.5 for each HPV type. Results: GMT ratios were 2.23, 3,17, 2.14, and 1.68 for types 6,11,16,& 18; Log transformed the data and calculated GMTs. Tested if post Dose 3 GMT ratio of the Alternate to Standard schedule was ≤ 0.5 for each HPV type

ADVERSE EVENTS:
Arm/Group | 6 Month Standard Schedule | 12 Month Alternative Group
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 57/100 | 55/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 Month Standard Schedule (N=100) | 12 Month Alternative Group (N=100)
Soreness at the injection site (Skin and subcutaneous tissue disorders) | 57 (114) | 55 (95)
syncope (General disorders) | 1 (1) | 0 (0) — One case of brief syncope in 6 month arm resolved without consequence.

LIMITATIONS AND CAVEATS:
One participant in the Standard group did not respond to any of the vaccine HPV types. Eleven participants in the Alternate group either did not receive Dose 3 or were out of window, compared with only one participant in the Standard group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less